CLINICAL TRIAL: NCT03368118
Title: A Follow-up Phase IIa Study to Evaluate the Long-term Safety and Efficacy Profile of ABX464 Given at 50 mg Once Daily in Subjects With Moderate to Severe Active Ulcerative Colitis.
Brief Title: Study Evaluating the Long-term Safety and Efficacy of ABX464 in Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX464-102
Record Dates: First submitted 2017-11-13; First posted 2017-12-11 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis
Keywords: ABX464; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ABX464

STUDY DESIGN:
Intervention Model Description: open-label, follow-up study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABX464 Treatment arm (Experimental): All subjects will receive ABX464 at 50 mg o.d for an overall period of 48 months.
  Interventions: Drug: ABX464

INTERVENTIONS:
Drug: ABX464 — All subjects will receive ABX464 given at 50 mg o.d for an overall period of 48 months.

SUMMARY:
This study is an open-label study aiming at evaluating the long-term safety and the efficacy profile of ABX464 given once a day (o.d) at 50 mg in subjects who have been previously enrolled in the ABX464-101 clinical study (induction study) and who are willing to continue their treatment.

DETAILED DESCRIPTION:
This study is an open-label study aiming at evaluating the long-term safety and the efficacy profile of ABX464 given once a day (o.d) at 50 mg in subjects who have been previously enrolled in the ABX464-101 clinical study (induction study) and who are willing to continue their treatment.

All subjects will receive ABX464 given at 50 mg o.d irrespective of their previous treatment received in the ABX464-101 study (i.e. ABX464 or Placebo).

The actual treatment received by a subject throughout the previous study (ABX464-101) will not be known at the time the subjects enter this follow-up study. This treatment group will be communicated (throughout the investigators) to the subjects at the end of the ABX464-101 study (planned in Q3/2018).

The enrolment in this follow-up study will be based on the willingness of the subject to carry on his/her participation and also based on investigator's judgement.

Subjects will be treated with ABX464 for an overall period of 48 months. Subjects will be followed up weekly during the first month, every two weeks during the second month and then on a monthly basis until M24, then quaterly from M24 to M48.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if ALL of the following criteria apply:

* Subjects previously enrolled in the ABX464-101 clinical study who have completed the initial 2-month treatment phase;
* Subjects able and willing to comply with study visits and procedures;
* Subjects with hematological and biochemical laboratory parameters as follows at the D56 visit of the ABX464-101 study:

  * Hemoglobin > 9.0 g dL-1;
  * Absolute neutrophil count ≥ 750 mm-3;
  * Platelets ≥ 100,000 mm-3;
  * Total serum creatinine ≤ 1.3 x ULN (upper limit of normal);
  * Creatinine clearance > 50 mL min-1 by the Cockcroft-Gault equation;
  * Total serum bilirubin < 1.5 x ULN;
  * Alkaline phosphatase, AST (SGOT) and ALT (SGPT) < 1.5 x ULN;
* Subjects should understand, sign and date the written voluntary informed consent form at the enrolment visit prior to any protocol-specific procedures being performed;
* Subjects should be affiliated to a social security regimen (for French sites only);
* Females and males receiving the study treatment and their partners must agree to use a highly effective contraceptive method during the study and for 3 months after end of study or early termination. Contraception should be in place at least 3 months prior to study participation. Women must be either postmenopausal (at least 12 months of amenorrhea), surgically sterile or if of childbearing potential must use a highly effective contraceptive method. Women of childbearing potential (WOCBP) will enter the study after confirmed menstrual period and a negative pregnancy test. Highly effective methods of contraception include: true abstinence, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), hormonal contraception (estrogen and progestogen or progestogen only) associated with inhibition of ovulation, bilateral tubal occlusion, vasectomized partner. True abstinence is defined when this is in line with the preferred and usual lifestyle of the subject. In each case of delayed menstrual period (over one month between menstruations) confirmation of absence of pregnancy is required. This recommendation also applies to WOCBP with infrequent or irregular menstrual cycle.

Exclusion Criteria:

The following criterion should be checked at the time of screening. If this exclusion criterion applies, the subject will not be included in the study:

▪ Any condition, which in the opinion of the investigator, could compromise the subject's safety or the adherence to the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul GINESTE, Study Director — Abivax S.A.
Locations (1):
- Department of Gastroenterology - University hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: preliminary results at M24 — https://www.abivax.com/press-releases/

RESULTS

PARTICIPANT FLOW:
Groups:
- ABX464 Treatment Arm: All subjects received ABX464 at 50 mg o.d for an overall period of 48 months.
  ABX464: All subjects received ABX464 given at 50 mg o.d for an overall period of 48 months.
Period: Overall Study
Arm/Group | ABX464 Treatment Arm
Started | 22
Completed | 11
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 3
  Poland | 10
  Hungary | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events
Description: Number of treatment-emergent adverse events in ABX464 treated subjects
Time Frame: Through subject study treatment, up to 48 months
Measure: Number; unit: events
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
events | 145

2. Secondary Outcome: Total Mayo Score
Description: The change from Day 0 up to Month 48 in Total Mayo Score. total mayo score is an index and consists of 4 items: stool frequency, rectal bleeding, flexible sigmoidoscopic examination, and a physician global assessment of disease activity.
  Each parameter of the score ranges from zero (normal or inactive disease) to 3 (severe activity). The total mayo score scale ranging is from 0 to 12 The change from baseline of this score is part of the clinical response definition: to get a clinical response, a reduction in Total Mayo score of at least 2 points is required. A higher (in negative) change shows a better clinical response.
Time Frame: Up to Month 48
Population: Non responder Imputation (NRI) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
units on a scale | -3.0 (3.4)

3. Secondary Outcome: Partial Mayo Score
Description: The change from Day 0 up to Month 48 in Partial Mayo Score; Partial Mayo score is an index and consists of 3 items: stool frequency, rectal bleeding and a physician global assessment of disease activity.
  Each parameter of the score ranges from zero (normal or inactive disease) to 3 (severe activity). The partial mayo score scale ranging is from 0 to 9.
  A higher (in negative) change from baseline shows a better clinical response
Time Frame: Up to Month 48
Population: Non responder imputation population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
units on a scale | -2.2 (2.4)

4. Secondary Outcome: Number of Subjects With Clinical Response at Month 48
Description: Clinical response was defined as:
  reduction in Total Mayo Score (TMS) of at least 2 points and >= 30 percent from baseline with an accompanying decrease in rectal bleeding sub-score of >= 1 point or absolute rectal bleeding sub-score of <= 1 point.
Time Frame: up to 48 months
Population: Non responder imputation population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
Participants | 11

5. Secondary Outcome: Number of Subjects With Clinical Remission at Month 48
Description: Clinical remission was achieved when all the following criteria were met in the components of the Mayo clinical Score:
  rectal bleeding sub-score = 0 central endoscopy sub-score <= 1 stool frequency sub-score <= 1
Time Frame: up to 48 months
Population: non responder imputation population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
Participants | 9

6. Secondary Outcome: Number of Subject With Endoscopic Improvement at Month 48
Description: oEndoscopic improvement was achieved if the Mayo central endoscopic sub-score is 0 or 1.
Time Frame: up to 48 Months
Population: Non responder imputation population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
Participants | 9

7. Secondary Outcome: Number of Subjects With Endoscopic Remission at Month 48
Description: Endoscopic remission was defined as Mayo central endoscopic sub-score = 0
Time Frame: up to 48 months
Population: non responder imputation population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
Participants | 6

8. Secondary Outcome: Fecal Calprotectin
Description: The change from Day 0 up to Month 48 in fecal calprotectin A higher (in negative) change shows a better efficacy
Time Frame: Up to Month 48
Population: Non responder imputation population
Measure: Mean (Standard Deviation); unit: ug/g
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
ug/g | -299.69 (472.28)

9. Secondary Outcome: CRP Levels
Description: The change from Day 0 up to Month 48 in CRP levels
Time Frame: Up to Month 48
Population: Non responder imputation population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
mg/L | 2.29 (4.82)

10. Secondary Outcome: Number of Treatment-emergent Serious Adverse Events
Description: The number of incidences of treatment-emergent serious adverse events
Time Frame: Through subject study treatment, up to 48 months
Population: Observed cases population
Measure: Number; unit: events
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
events | 3

11. Secondary Outcome: Number of Treatment-emergent Adverse Events of Special Interest
Description: The number of incidences of treatment-emergent adverse events of special interest
Time Frame: Through subject study treatment, up to 48 months
Population: Observed cases population
Measure: Number; unit: events
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
events | 15

12. Secondary Outcome: Number of Adverse Events Leading to Investigational Product Discontinuation
Description: The number of incidences of adverse events leading to investigational product discontinuation
Time Frame: Through subject study treatment, up to 48 months
Population: Observed cases population
Measure: Number; unit: event
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
event | 1

13. Secondary Outcome: Number of Specific Laboratory Abnormalities
Description: The number of incidences of specific laboratory abnormalities
Time Frame: Through first year of subject study treatment, 12 months
Population: Observed Cases
Measure: Number; unit: events
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
events | 17

14. Secondary Outcome: SF-36 Quality of Life Questionnaire (SF-36 Physical Component)
Description: Change from Day 0 up to 24 months in SF-36 Questionnaire scores; The SF-36 questionnaire is a self-administered questionnaire containing 36 items.
  It measures health on eight multi-item dimensions, covering functional status, well-being, and overall evaluation of health.
  These items are grouped in 2 distincts components: a physical component (SF-36 physical) and a mental component (SF-36 mental).
  This outcome describes the SF-36 physical component. Each item score ranging is from 0 to 100. A higher positive value in change indicate a better health status. The higher the change from baseline, the better improvement
Time Frame: Up to 24 months
Population: Non responder imputation population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
units on a scale | 4.82 (4.23)

15. Secondary Outcome: SF-36 Quality of Life Questionnaire (SF-36 Mental Component)
Description: Change from Day 0 up to 24 months in SF-36 Questionnaire scores; The SF-36 questionnaire is a self-administered questionnaire containing 36 items.
  It measures health on eight multi-item dimensions, covering functional status, well-being, and overall evaluation of health.
  These items are grouped in 2 distincts components: a physical component (SF-36 physical) and a mental component (SF-36 mental).
  This outcome describes the SF-36 mental component. Each item score ranging is from 0 to 100. A higher positive value in change indicate a better health status. The higher the change from baseline, the better improvement
Time Frame: Up to 24 months
Population: Non responder imputation population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
units on a scale | 6.38 (3.40)

16. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) Levels
Description: The change from Day 0 up to Month 48 in ESR levels
Time Frame: up to 48 Months
Population: Non responder imputation population
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
mm/hour | 2.90 (8.62)

17. Post Hoc Outcome: UC Worsening
Description: Proportion of subjects with UC worsening based on adverse events
Time Frame: Up to Month 48
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 Treatment Arm
Number analyzed (Participants) | 22
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse event were collected from first day of dosing (baseline) up to last safety visit (up to 49 months : 48 months on treatment and one month safety follow-up)
Arm/Group | ABX464 Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 Treatment Arm (N=22)
Myocardial infarction (Cardiac disorders) | 1 (1) — The event was considered not related to study treatment and resolved without sequelae 5 days after onset date. No action was taken with study treatment
enteropathic spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) — The subject admitted to hospital due to spondyloarthropathy caused by inflammatory bowel disease (HLA-B27+). The event considered not related to study treatment and resolved without sequelae. No action was taken with study treatment.
benign ovarian tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — subject underwent total hysterectomy. Event considered not related to study treatment and resolved without sequelae. Study treatment was temporarily discontinued.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 Treatment Arm (N=22)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
colitis ulcerative (Gastrointestinal disorders) | 7 (11)
diarrhoea (Gastrointestinal disorders) | 4 (10)
Dyspepsia (Gastrointestinal disorders) | 2 (3)
nausea (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 3 (4)
Pyrexia (General disorders) | 2 (2)
nasopharyngitis (Infections and infestations) | 5 (9)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
headache (Nervous system disorders) | 3 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT03368118/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT03368118/SAP_001.pdf